CLINICAL TRIAL: NCT01937195
Title: A Prospective, Randomized, Controlled, Multicenter Comparison Between the AccuCath™ Intravenous Catheter System With Retractable Coiled Tip Guidewire and Conventional Peripheral Intravenous Catheters With a Vascular Access Team
Brief Title: AccuCath™ Intravenous (IV) Device Used by Vascular Access Team (VAT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VPW-STP-00002
Record Dates: First submitted 2013-04-15; First posted 2013-09-09 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-03

CONDITIONS: Vascular Access Complication
Keywords: IV Catheter comparison; AccuCath versus Conventional IV Catheters; IV Catheter Study; IV Catheter User Preference Comparison; First Attempt Success Rate for IV Catheters; AccuCath Device Performance; Complication Rates for IV Catheters; Average Dwell Time for IV Catheters; Patient Satisfaction with IV Catheters; Clinician Satisfaction with AccuCath Device Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AccuCath Intravenous Catheter System (Experimental): AccuCath Intravenous Catheter System will be used for IV therapy during inpatient stay. Intervention includes vascular access, fluid infusion, and blood sample removal.
  Interventions: Device: AccuCath Intravenous Catheter System

INTERVENTIONS:
Device: AccuCath Intravenous Catheter System — AccuCath IV Catheter System will be used for IV therapy during inpatient stay. Intervention includes vascular access, fluid infusion, and blood sample removal. Results will be compared to published literature for conventional IV catheters.

SUMMARY:
The study will test a hypothesis that the AccuCath™ System will have a higher rate of successful first attempt peripheral intravenous (PIV) placement, higher completion of therapy, fewer complications, longer dwell times, and higher user satisfaction compared to Conventional IV Catheters.

DETAILED DESCRIPTION:
Phase One is designed as a one-arm prospective study to compare patients using the AccuCath™ Intravenous Catheter System to the results found in literature. Phase Two is designed as a two-arm prospective randomized controlled study comparing the AccuCath™ Intravenous Catheter System to conventional PIV catheters. This study site will be completing Phase One only.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age > or equal to 18 years or < or equal to 89 years old;
2. Capable and willing to give informed consent;
3. English speaking;
4. Acceptable candidate for an elective, non-emergent PIV as determined by ordering physician;
5. Admitted to study inpatient unit.

Exclusion Criteria:

1. Male or female, < 18 years old or > 89 years old;
2. Requirement for emergent IV placement (patient's condition would be compromised if there is a delay in IV placement);
3. Previous venous grafts or surgery at the target vessel access site;
4. Currently involved in other investigational clinical trials (unless permission is granted by other study PI);
5. Females who are pregnant, planning to become pregnant within 3 months of the procedure, or lactating.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman R Anderson, RN, Principal Investigator — Evangelical Community Hospital
Locations (1):
- Evangelical Community Hospital, Lewisburg, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Anderson NR. Influencing Patient Satisfaction Scores: Prospective One-Arm Study of a Novel Intravenous Catheter System With Retractable Coiled-Tip Guidewire Compared With Published Literature for Conventional Peripheral Intravenous Catheters. J Infus Nurs. 2016 Jul-Aug;39(4):201-9. doi: 10.1097/NAN.0000000000000173. PMID 27379678

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from April 2013 through June 2014. Patients were admitted to the inpatient units at Evangelical Community Hospital.
Groups:
- AccuCath Intravenous Catheter Device: AccuCath Intravenous Catheter System: AccuCath IV Catheter System (study device) will be used for IV therapy during inpatient stay. Intervention includes vascular access, fluid infusion, and blood sample removal. Results will be compared to published literature for conventional IV catheters.
Period: Overall Study
Arm/Group | AccuCath Intravenous Catheter Device
Started | 95
Completed | 95
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Inpatients requiring IV therapy during hospital admission of > 24 hours.
Arm/Group | AccuCath Intravenous Catheter Device
Number analyzed (Participants) | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 95
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 95

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Successfully Inserted Peripheral IV Catheter Placement on First Attempt
Description: The primary endpoint is to observe the rate of first attempt success (where the inserter only pierces the skin once and successfully places the PIV catheter in the vein) in patients requiring PIV access.
Time Frame: Baseline/at catheter placement, usually 3-15 minutes initial during insertion procedure
Population: Inpatients requiring IV therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AccuCath Intravenous Catheter Device
Number analyzed (Participants) | 95
percentage of participants | 85.3 [76.5 to 91.7]

2. Secondary Outcome: Percentage of Patients With Complications of Peripheral IV Therapy
Description: Will measure the percentage of patients with (anticipated) complications of IV therapy - infection, occlusion, infiltration, extravasation, phlebitis, dislodgement, leaking/bleeding at site, patient complaints of pain without other identifiable cause, and other (up to 7 days).
Time Frame: Study exit/at catheter removal expected to be up to 7 days post placement
Population: Inpatient units requiring IV therapy.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | AccuCath Intravenous Catheter Device
Number analyzed (Participants) | 95
percentage of patients | 17.9 [10.8 to 27.1]

3. Secondary Outcome: Completion of IV Therapy
Description: Completion of IV therapy will measure whether the catheter remained in place for the duration of required intravenous treatment during the inpatient stay (generally up to 7 days).
Time Frame: Study exit/at catheter removal expected to be up to 7 days post placement
Population: Inpatients requiring IV therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | AccuCath Intravenous Catheter Device
Number analyzed (Participants) | 95
Participants | 78

4. Secondary Outcome: Catheter Dwell Time
Description: Will measure total catheter dwell time to the nearest hour (total time in hours for functioning catheter) up to 7 days.
Time Frame: Study exit/at catheter removal expected to be up to 7 days post placement
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | AccuCath Intravenous Catheter Device
Number analyzed (Participants) | 95
hours | 58 [49.1 to 66.8]

5. Secondary Outcome: Percentage of Patients Who Identified as "Satisfied" With Catheter Performance at Catheter Insertion
Description: Patients were surveyed regarding satisfaction with catheter insertion with a 5-point Likert scale (1 the lowest, 5 the highest). Satisfaction was defined as a score of 3 to 5.
Time Frame: Baseline at catheter insertion in the first 3-15 minutes after procedure
Population: Inpatients requiring IV therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AccuCath Intravenous Catheter Device
Number analyzed (Participants) | 95
percentage of participants | 100.0 [96.2 to 100]

6. Secondary Outcome: Number of Participants Experiencing Adverse Events
Description: Will measure the number and severity of adverse events associated with peripheral IV initiation and indwelling catheter time up to 7 days. Adverse events are anticipated complications of IV therapy.
Time Frame: baseline, and up to catheter removal expected to be no more than 7 days post placement
Population: Inpatients requiring IV therapy.
Measure: Number; unit: participants
Arm/Group | AccuCath Intravenous Catheter Device
Number analyzed (Participants) | 95
participants
  Total | 17
  Phlebitis | 7
  Infiltration | 6
  Leaking | 3
  Dislodgement | 1

7. Secondary Outcome: Percentage of Patients Who Identified as "Satisfied" With Catheter Performance at Catheter Removal
Description: Patients were surveyed regarding satisfaction with catheter performance with a 5-point Likert scale (1 the lowest, 5 the highest). Satisfaction was defined as a score of 3 to 5.
Time Frame: At catheter removal, which is expected to be up to 7 days post placement
Population: Inpatients requiring IV therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AccuCath Intravenous Catheter Device
Number analyzed (Participants) | 95
percentage of participants | 97.9 [92.6 to 99.7]

ADVERSE EVENTS:
Time Frame: During enrollment from April 2013 through June 2014.
Description: IV complications are anticipated events during conventional IV therapy and occur about 47% of the time.
Arm/Group | AccuCath Intravenous Catheter Device
Serious Adverse Events (participants affected / at risk) | 0/95
Other Adverse Events (participants affected / at risk) | 17/95
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AccuCath Intravenous Catheter Device (N=95)
Vascular Complication (Vascular disorders) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No